CLINICAL TRIAL: NCT00839267
Title: The Comparison of Clopidogrel Efficacy in Patients With Acute Myocardial Infarction and Severe Hemodynamic Instability to Patients With Hemodynamically Uncomplicated Myocardial Infarction
Brief Title: Clopidogrel Efficacy and Acute Coronary Syndromes
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Pavel Osmancik, Charles University Prague
Other Study IDs: CLO-OSM-02
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Acute Myocardial Infarction
Keywords: platelet; VASP; clopidogrel; cardiogenic shock; myocardial infarction; percutaneous coronary intervention
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Unstable: Patient with acute myocardial infarction plus severe hemodynamical instability. It means, on mechanical ventilation and catecholamine support
- Stable: Patients with myocardial infarction hemodynamically completely (Killip I)stable.

SUMMARY:
The purpose of this study is to compare clopidogrel effectiveness between severe hemodynamically unstable versus stable patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Clopidogrel exists in oral form only. As a prodrug, it has to be metabolized to the active form by cytochrome system in the liver. Both facts could lead to lower efficacy of the drug in hemodynamically unstable patients, where splanchnic and liver hypoperfusion is present. We hypothesised that clopidogrel efficacy is insufficient in patients with acute myocardial infarction and severe hemodynamic instability. Therefore we would like to compare the effect of clopidogrel in unstable STEMI patients on mechanical ventilation with stable STEMI patients.

ELIGIBILITY:
Inclusion Criteria for unstable group:

* acute STEMI
* mechanical ventilation
* the need for catecholamine support.

Inclusion Criteria for stable group:

* acute myocardial infarction

Exclusion Criteria for any:

* previous treatment with clopidogrel
* clopidogrel administration during transport by ambulance
* known intolerance to clopidogrel
* history of thrombocytopenia (<150,000 platelets/ml)
* pre-existing liver disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of 40 consecutive patients is planned, all of them with acute myocardial infarction with ST-segment elevation.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-06; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Lower efficacy of clopidogrel determined by VASP measurement | 6 months

SECONDARY OUTCOMES:
Higher frequency of stent thrombosis in the unstable group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Osmancik, MD, PhD, Principal Investigator — Charles University Prague
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia